CLINICAL TRIAL: NCT05167331
Title: Efficacy of Virtual Reality Hypnosis Versus Nitrous Oxide Inhalation on Children's Anxiety During a Dental Treatment : a Randomized Clinical Trial
Brief Title: Comparative Clinical Study Between Virtual Reality Hypnosis and Nitrous Oxide Inhalation for Dental Anxie
Acronym: HYPNOSEDENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8113
Record Dates: First submitted 2021-11-25; First posted 2021-12-22 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Dental Anxiety
Keywords: virtual reality; hypnosis; nitrous oxide; dental anxiety; child

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Active Comparator): * (T1) after fitting the headset to the child's face, the assistant starts the VR program chosen by the child.
  * (T2) Five minutes after induction, local anesthesia with the QUICKSLEEPER device is performed. The injection of a cartridge of anesthetic Articaïne SEPTANEST 1/200 000 is administered intraosseously.
  * (T3) After placing the rubber dam, the investigator performs restorative +/- endodontic care of the selected temporary molar.
  * (T4) Once the treatment is finished, the sedation is stopped and the patient rests in the chair for 5 minutes.
  * (T5) As soon as the investigator considers that the child is back to normal state, he can leave the office with his parents.
  Interventions: Device: Dispositif de RV - HYPNO VR
- Nitrous oxide sedation (Active Comparator): * (T1) With the nitrous oxide/oxygen inhalation system titrated to 50%/50% whose flow rate is adapted to the child's respiratory flow. The assistant is responsible for controlling the sedation. Verbal encouragement is always present to reassure the child.
  * (T2) Five minutes after induction, local anesthesia with the QUICKSLEEPER device is performed. The injection of a cartridge of anesthetic Articaïne SEPTANEST 1/200 000 is administered intraosseously.
  * (T3) After placing the rubber dam, the investigator performs restorative +/- endodontic care of the selected temporary molar.
  * (T4) Once the treatment is finished, the sedation is stopped and the patient rests in the chair for 5 minutes.
  * (T5) As soon as the investigator considers that the child is back to normal state, he can leave the office with his parents.
  Interventions: Drug: Nitrous Oxide inhalation

INTERVENTIONS:
Drug: Nitrous Oxide inhalation — use of Nitrous Oxide inhalation on children's anxiety during a dental treatment
  Arms: Nitrous oxide sedation
Device: Dispositif de RV - HYPNO VR — use of Virtual Reality on children's anxiety during a dental treatment
  Arms: Virtual Reality

SUMMARY:
The vicious circle of dental anxiety impacts major aspects of a child's quality of life. Hypnosis using distraction is one of the most common non-pharmalogical techniques in behavior and pain management in pediatric dentistry. Its value over traditional pharmalogical sedation is undeniable. This clinical study examines the application of hypnosis delivered through immersive virtual reality (VR) for anxious children ongoing dental procedures. The investigators will explore whether VR is as effective on pain and anxiety relief as a pharmacological sedation with inhalation of nitrous oxide.

DETAILED DESCRIPTION:
The working hypothesis of this study is that hypnosis through virtual reality can reduce children's anxiety as well as their pain level during dental care with an efficiency and tolerance at least similar to nitrous oxide inhalation. Specifically, the statistical analyses will be based on an assumption of non-inferiority of VR compared to the pharmacological technique of nitrous oxide sedation.

Each patient (aged from 6 to 10) attended for two visits in order to benefit of 2 similar conservative dental treatments on primary molars.

Everyone was randomly allocated to receive hypnosis through virtual reality or nitrous oxide/oxygen titrated to 50%/50% at the first visit, the alternative being used at the second visit. This randomization helps avoid any experimental bias related to a first positive or negative experience, each patient being its own control.

Vital signs and a video of the child's behavior are recorded for an external examinator. The video shows the child's body response as an indicator for his anxiety level through the procedures. The child's face doesn't appear on the video in order to reduce risks of bias.

ELIGIBILITY:
Inclusion criteria:

* Patients aged between 7 and 10 years
* With an indication for conservative and/or endodontic care of at least 2 temporary molars belonging to the same dental arch, unilateral or bilateral, and equivalent in terms of caries and symptoms
* With dental anxiety
* ASA I patients

Exclusion criteria:

* Patient with a history of MEOPA or virtual reality sedation for dental treatment
* Patient refusing to do preoperative intra-oral x-rays
* Patient with one of the MEOPA contraindications
* Patient with a history of post-operative nausea vomiting or motion sickness
* Patient with visual or hearing disorders
* Patient presenting with a psychiatric pathology or having taken psychotropic drugs in the 8 weeks preceding the 1st visit and during the duration of the study
* Patient with claustrophobia
* Patient without French Social Security coverage
* Lack of consent from the holders of parental authority to participate in the study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Anxiolysis assessed by a standardized hetero-assessment scale (Venham Modified Scale) | 5 weeks
  Child behavior can be assessed using the Veerkamp Modified Venham Scale (VMS). This is a scale from 0 (completely calm and relaxed patient) to 5 (distressed patient, completely disconnected). Several parameters are taken into account in this scale such as: the child's movements, crying or screaming, the possibility or not of performing the treatment. The authors have found this scale to be a reliable, easy-to-use and reproducible instrument when it comes to assessing children's behavior.
  This outcome measure is assessed by an external examinator with the video recording the procedures.

SECONDARY OUTCOMES:
Assessment of analgesia with VR | 5 weeks
  Assessment of analgesia using self-assessed pain levels on standardized age-appropriate scales (VAS: Visual Analogue Scale)
Assessment of children's tolerance levels to VR and pharmacological technique. | 5 weeks
  Assessment of tolerance and response to VR-MEOPA using the number and proportion of patients intolerant to VR and to pharmacological techniques. Evaluate the proportion of VR or MEOPA sessions interrupted (lack of therapeutic continuity). Any patient who has interrupted VR more than once or who refused VR during the procedure is considered intolerant of VR.
Assessment of the impact of the child's temperament on his acceptance of nitrous oxide and RV sedations using a questionnaire and a temperament scale | The parents answer to the questionnaire on the first visit during inclusion.
  To assess the child's temperament dimensions, parents answer to an Emotionality, Activity and Sociability questionnaire with the help of an investigator before the treatment session. The AES questionnaire had already been validated in France in children aged from 6 to 12 years-old in 2002. The AES questionnaire is a questionnaire containing 25 items based on a model of three main dimensions: Emotionality, Activity and Sociability. Each item has a Likert-type scale ranging from 1 (extremely false, not at all corresponding to my child) to 5 (extremely fair, corresponding to my child).

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Do NM, Maniere MC, Lefebvre F, Clauss F. Efficacy of virtual reality hypnosis versus conscious sedation with nitrous oxide in the management of dental anxiety in pediatric dentistry: protocol for a prospective randomized controlled trial. Trials. 2025 Jun 9;26(1):201. doi: 10.1186/s13063-025-08849-z. PMID 40490788